CLINICAL TRIAL: NCT04337476
Title: The Effects of Pacifier Activated Lullaby in VLBW Preterm Infants: an Italian Randomized Pilot Study
Brief Title: The Effects of Pacifier Activated Lullaby in VLBW Preterm Infants
Acronym: PAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Barbara Sgobbi, Music Therapist, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAL- 176
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Music Therapy
Keywords: Music therapy; Preterm; PAL; HRV; Parental voice
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial, divided into four parallel groups of preterm infants
Who Masked: Care Provider, Investigator
Masking Description: After acquiring informed consent, participants will be randomized randomly through computerized, block randomization by intervention group or group of control, which will assign a specific group to the newborns (mom voice, dad voice, music therapist voice or no voice). The clinical team and parents will be blind to the study group and will not know when the recordings will be reproduced. The administration of the PAL and the reproduction of the relative voices will be performed by the music therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mother's song (Experimental): At the suggestion of the music therapist, the mothers of each child will record two lullabies sung by themselves; lullabies will be part of traditional classical literature. The songs will be recorded and loaded on a simplified digital software to modify any background noise or pauses. The recording will be inserted in the usb / sd flash drive used directly by the PAL device. During the entire hospital stay, newborn babies will receive standard care in use in the neonatal intensive care unit
  Interventions: Device: The effects of Pacifier Activated Lullaby in very low birth weigt preterm infants. An italian music therapy intervention
- father's song (Experimental): At the suggestion of the music therapist, the fathers of each child will record two lullabies sung by themselves; lullabies will be part of traditional classical literature. The songs will be recorded and loaded on a simplified digital software to modify any background noise or pauses. The recording will be inserted in the usb / sd flash drive used directly by the PAL device. During the entire hospital stay, newborn babies will receive standard care in use in the neonatal intensive care unit
  Interventions: Device: The effects of Pacifier Activated Lullaby in very low birth weigt preterm infants. An italian music therapy intervention
- singing of the music therapist (Experimental): Music therapist will record two lullabies sung by themselves; lullabies will be part of traditional classical literature. The songs will be recorded and loaded on a simplified digital software to modify any background noise or pauses. The recording will be inserted in the usb / sd flash drive used directly by the PAL device. During the entire hospital stay, newborn babies will receive standard care in use in the neonatal intensive care unit
  Interventions: Device: The effects of Pacifier Activated Lullaby in very low birth weigt preterm infants. An italian music therapy intervention
- No singing (No Intervention): Control group (not subjected to musical stimulation- no singing). During the entire hospital stay, newborn babies will receive standard care in use in the neonatal intensive care unit.

INTERVENTIONS:
Device: The effects of Pacifier Activated Lullaby in very low birth weigt preterm infants. An italian music therapy intervention — Positive reinforcement is an effective development strategy for improving the feeding skills of preterm infants. A brief intervention with the PAL device with pacifier that reproduces lullabies sung by both parents or by the music therapist could reduce the use of the feeding tube and the length of hospital stay in preterm infants. The aim of this study is not only to evaluate the benefits of positive reinforcement on the nutritional sucking competence of the premature baby, but at the same time to observe its possible effects on its well-being and its clinical stability.
  Arms: father's song; mother's song; singing of the music therapist

SUMMARY:
Music and music therapy, live or recorded, has been introduced in the Neonatal Intensive Care Unit (NICU) of the Del Ponte hospital in Varese in addition to standard medical and nursing care, to improve premature neonates' neurophysiological development.

Recent studies focused on the effects of the maternal voice or the entrained singing and live music, highlighting their benefits on neonates stress, on not-nutritive sucking and on the caloric intake.

Aim of our study is to evaluate the effect of parents singing or musictherapist singing admistered by Pacifier Activated Lullaby (PAL) on infant's behavior and nutritional outcomes.

Particularly, we will evaluate infants' Heart Rate Variability during music therapy session, exclusive oral feeding achievement, weigth increase and hospitalization in a group of preterm infants administered to PAL compared with a control group of preterm infants not exposed to PAL stimulus.

DETAILED DESCRIPTION:
A Prospective randomized controlled pilot study trial will be conducted. Infants will be evaluated at 32-34 post-conceptional weeks when the volume of milk assumed orally will be less than 50% of the total enteral intake.

Infants with gestational age less than 34 weeks will be enrolled. After the request for informed consent, participants will be randomized randomly through computerized.

The administration of the PAL and the reproduction of the relative voices will be performed by the music therapist.

Objective of this study is to evaluate the tolerance (in terms of clinical stability, described through the HRV parameter) of the PAL device by the enrolled customers and investigate any benefits of the positive reinforcement purchased, through its use, on the acquisition of food skills and on the growth of preterms.

Primary Outcome: Clinical Stability Using Heart Rate Variability (HRV) Measurement during the music therapy treatment.

Secondary Outcomes: effects of positive reinforcement (obtained through the use of the device PAL) on the acquisition of food skills and the growth of preterm consumers.

In particular:

* Evaluation of the achievement of the exclusive oral sucking
* Evaluation of the variation in the rate of meal intake between the beginning and the end of the intervention
* Assessment of the infant's weight gain in the 24 hours following stimulation
* Evaluation of the rate of growth from the last day of treatment to discharge.
* Duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between the 23th and the 34th week, sufficient stability of the vital parameters and absence of active infections and episodes of apnoea during the 72 hours before the test

Exclusion Criteria:

* Chromosomal aberrations, congenital maxillofacial malformations, respiratory support at evaluation time Neonates with failed responses to bilateral hearing screening performed by Automated Auditory Brainstem Response testing will be subsequently excluded

Infants will be evaluated at 32-34 post-conceptional weeks when the volume of milk assumed orally will be less than 50% of the total enteral intake

Ages: 23 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | through study completion (from 5 minutes before the test to 5 minutes after the test ended)
  Heart Rate Variability (HRV) according to different music genres listening. An electrocardiogram is performed to evaluate HRV parameters during the test's administration

SECONDARY OUTCOMES:
Full oral feeding | more or less than 35 post conceptional weeks
  Full oral feeding (> 150 ml/kg/day) achievement, expressed as post-conceptional weeks.
oral feeding velocity | more or less than 30 minutes
  time (expressed as minutes) necessary to consume oral feeding
weight gain | 24 hours after test
  % weight increase 24 hours after test administration
lenght of stay | more or less than 36 post conceptional weeks
  length of hospitalization (expressed as post-conceptional weeks at discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Agosti, MD, Principal Investigator — Neonatologia, TIN e Pediatria Verbano- Ospedale F. del Ponte
Locations (1):
- Ospedale F. Del Ponte, Varese, Italy

IPD SHARING:
Plan to Share IPD: No